CLINICAL TRIAL: NCT04542044
Title: Evaluation of the Safety and Outcomes of Outpatient Management With Mild to Moderate COVID-19 Pneumonia (PneumoCoV-Ambu)
Brief Title: Evaluation of the Safety and Outcomes of Outpatient Management With Mild to Moderate COVID-19 Pneumonia
Acronym: PneumoCoV-Ambu
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Chevallier-Lugon Chloé, Chief resident, University Hospital, Geneva
Other Study IDs: CCER2020-01518
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: management strategy of outpatient with mild to moderate SARS-CoV-2 pneumonia — Data collected with a cohorte of SARS-CoV-2 pneumonia in an outpatient basis

SUMMARY:
The purpose of this study is to evaluate the strategy of investigators for outpatients SARS-CoV-2 moderate pneumonia management in terms of efficacy and patient safety. The investigators ultimate goal is to validate first wave management strategy in order to support the investigators future approach in the event of a second wave, and spare the hospital resources by safely keeping at home as many patients as possible.

DETAILED DESCRIPTION:
The investigators focused on participants consulting in the emergency department at the HUG who remained in an outpatient setting, with pneumonia and moderate illness, defined by individuals who have evidence of lower respiratory disease by clinical assessment or imaging and a saturation of oxygen (SaO2) >93% on room air and no other hospitalization criteria (CURB 65 score below 2points).

For patients' follow-up, the investigators have created an aftercare ambulatory unit, open 5/7 days. The investigators were able to conduct 64 consultations between April 2 and May 5, 2020. Every participant had suspected or confirmed SARS-CoV-2 pulmonary tract infection.

The follow-up data was entered into DPI (patient's medical record at HUG) on a specific consultation form. Patients followed in the investigators consultation were contacted between 30 and 60 days after diagnosis by the Covicare team. The Covicare team is call-center composed of medical students and primary care physicians who remotely followed patients with COVID-19 by calling them by phone or telemedicine every day or every other day depending on patients' needs and health status. The investigators will export data from RedCap concerning post-hospitalization, satisfaction survey on our care and oral consent for use of data (ARGOS study CCER number 2020-01273).

ELIGIBILITY:
Inclusion Criteria:

* All persons with suspected or confirmed SARS-CoV-2 pneumonia who consulted in the emergency department of the HUG without criteria for hospitalization4 (Pneumonia with CURB-65 >= 2 or new O2 dependency or increased O2 requirements or sustained respiratory rate≥20 min or decompensated comorbidity or major alteration of the general state) and who have been scheduled for outpatient follow-up in HUG.

Exclusion Criteria:

* Patients with hospitalization criteria
* Refusal to consent documentation found in the computerized patient record or oral refusal consent during follow up call.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with SARS-CoV-2 pneumonia without hospitalization criteria at primary consultation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Secondary hospitalization(s) or death COVID-19 related | 30 to 60 days from diagnosis

SECONDARY OUTCOMES:
severity of COVID-19 disease | 30 to 60 days from diagnosis
  severity of COVID-19 disease on a 7-points ordinal scale (1: not hospitalized, no limitation of activities; 2: not hospitalized, limitation of activities; 3: hospitalized, not requiring supplementary oxygen; 4: hospitalized, requiring supplementary oxygen; 5: hospitalized, on non-invasive mechanical ventilation; 6: hospitalized, on invasive mechanical ventilation or ECMO; 7: death),
patient satisfaction with management strategies | 30 to 60 days from diagnosis
  Satisfaction Survey of outpatient management
Saved costs | 30 days
  estimation of saved costs compared with a strategy of hospitalization of all COVID-19 related pneumonia cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT04542044/Prot_000.pdf